CLINICAL TRIAL: NCT03107780
Title: Phase 0/I Study of AMG 232 (KRT 232) Concentrations in Brain Tissue in Patients With Recurrent Glioblastoma and of AMG 232 (KRT 232) in Combination With Radiation in Patients With Newly Diagnosed Glioblastoma and Unmethylated MGMT Promoters
Brief Title: Testing the Ability of AMG 232 (KRT 232) to Get Into the Tumor in Patients With Brain Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00568; NCI-2017-00568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALLIANCE-ABTC-1604; ABTC-1604 (Other: Alliance for Clinical Trials in Oncology); ABTC-1604 (Other: CTEP); U10CA180821 (NIH); UM1CA137443 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma; Gliosarcoma; MGMT-Unmethylated Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (MDM2 inhibitor AMG 232 [KRT-232]) (Experimental): See Detailed Description
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Drug: Navtemadlin; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Navtemadlin — Given PO
  Other Names: (3R,5R,6S)-5-(3-Chlorophenyl)-6-(4-chlorophenyl)-3-methyl-1-((1S)-2-methyl-1-(((1-methylethyl)sulfonyl)methyl)propyl)-2-oxo-3-piperidineacetic Acid; AMG 232; AMG-232; KRT 232; KRT-232; KRT232; MDM2 Inhibitor KRT-232
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of navtemadlin in treating patients with glioblastoma (brain cancer) that is newly diagnosed or has come back (recurrent). Navtemadlin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the concentration and variability in concentration of navtemadlin (AMG 232 [KRT 232]) in brain and brain-associated tissue in patients with recurrent glioblastoma (GBM). (Part 1) II. Determine the maximum tolerated dose (MTD) of AMG 232 (KRT 232) given in combination with standard radiation following surgery for patients with newly diagnosed GBM harboring unmethylated MGMT promoters and wild-type TP53. (Part 2)

SECONDARY OBJECTIVES:

I. Determine the safety and toxicity of AMG 232 (KRT 232) in patients with recurrent GBM. (Part 1) II. Assess the variability of AMG 232 (KRT 232) concentration in tumor enhancing versus (vs.) infiltrative tissue. (Part 1) III. Assess the pharmacodynamic effect of AMG 232 (KRT 232) on p21 elevation. (Part 1) IV. Determine the safety of AMG 232 (KRT 232) given concurrently with radiation therapy (RT) and adjuvantly as monotherapy for patients with newly diagnosed GBM harboring unmethylated MGMT promoters and wild-type TP53. (Part 2) V. Assess AMG 232 (KRT 232) exposure and correlations with pharmacodynamic (PD) effect on p21 elevation. (Part 2) VI. Assess PD effect on MIC-1 elevation in serum. (Part 2)

OUTLINE: This is a phase 0, intratumoral pharmacokinetic (PK)/PD study of navtemadlin followed by a phase I dose-escalation study.

PART I: Patients with recurrent glioblastoma receive navtemadlin (KRT-232) orally (PO) once daily (QD) for 2 days. Within 3-6 hours of the last dose, patients undergo standard-of-care surgery. Upon recovery (within 45 days), patients with TP53 wild-type tumors continue to receive navtemadlin (KRT-232) PO QD on days 1-7. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) at baseline as well as on study and/or end of treatment and collection of blood and tissue samples at baseline and on study.

PART II: Within 6 weeks of standard-of-care surgery, patients with newly diagnosed glioblastoma undergo radiation therapy daily during weeks 1-6. Patients also receive navtemadlin (KRT-232) PO 1 time weekly (day 2), 2 times weekly (days 2, 4), 3 times weekly (days 2, 3, 5), 4 times weekly (days 2, 3, 4, 5), or 5 times weekly (days 1-5) for 6 weeks during radiation therapy. Patients also undergo MRI at baseline and end of treatment and collection of blood samples at baseline and on study.

PART II (EXPANSION COHORT): Patients receive navtemadlin (KRT-232) PO QD on days 1-7. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI at baseline, on study, and end of treatment.

After completion of study treatment, patients are followed every 2 months for the first two years from the off-treatment date, and then every 6 months until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Hemoglobin >= 10 g/dL (transfuse as necessary to raise levels, no transfusions within 7 days of start)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Alkaline phosphatase < 2.0 x ULN
* Creatinine =< institutional ULN
* Creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Patients must be able to provide written informed consent
* Patients must have MRI within 21 days before starting treatment; patients must be able to tolerate MRI with gadolinium
* Patients must be maintained on a stable corticosteroid regimen (no increase for 5 days) prior to the baseline MRI
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation through 5 weeks (women) after receiving the last dose of AMG 232 (KRT 232); should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of AMG 232 (KRT 232) administration; adequate methods of effective birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or intrauterine device (IUD) (women); bilateral tubal ligation (women)
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must be able to swallow oral medications
* PART 1 PATIENTS (SURGICALLY ELIGIBLE RECURRENT GBM)
* Part 1 patients must have prior histologically proven glioblastoma that is progressive or recurrent following radiation therapy +/- chemotherapy
* Part 1 patients must be undergoing repeat surgery that is clinically indicated as determined by their care providers
* Part 1 patients must have a tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of glioblastoma completed and signed by a pathologist
* Part 1 patients may have an unlimited number of prior therapy regimens
* Part 1 patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy or mitomycin C
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent, except bevacizumab/VEGFR inhibitors (e.g., erlotinib, hydroxychloroquine, etc.)
  * 6 weeks from bevacizumab/VEGFR inhibitors
* PART 2 PATIENTS (NEWLY DIAGNOSED GBM)
* Part 2 patients must have histologically confirmed glioblastoma or gliosarcoma
* Part 2 patients must have recovered from the immediate post-operative period
* Part 2 patients must have tumor MGMT methylation status of unmethylated; results of routinely used methods for MGMT methylation testing (e.g. mutagenically separated polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable
* Part 2 patient must show evidence of wild-type (WT) p53 status on somatic tissue specimens as assessed by deoxyribonucleic acid (DNA) sequencing
* Part 2 patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor infiltrating lymphocytes [TIL], LAK or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Part 1 patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are ineligible
* Patients with a history of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to AMG 232 (KRT 232) are ineligible; the AMG 232 (KRT 232) investigator brochure can be referenced for more information
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of AMG 232 (KRT 232)
* Patients may not use herbal or non-traditional medications while receiving AMG 232 (KRT 232) therapy; all herbal medicines (e.g., St. John's wort), and supplements consumed by the subject within the 30 days prior to receiving the first dose of AMG 232 (KRT 232) should be reviewed by the principal investigator
* Drugs known to be sensitive CYP3A4 substrates with narrow therapeutic windows (such as alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, sirolimus, or terfenadine) are not allowed; patients must be switched to alternative drugs at least 14 days prior to receiving the first dose of AMG 232 (KRT 232); those patients who cannot switch to alternative drugs will be excluded from the study; please note that the list of drugs above is not an exhaustive list; refer to reliable sources such as the FDA website (Drug development and drug interactions), or Micromedex when evaluating potential drug-interactions
* Treatment with medications known to cause corrected QT (QTc) interval prolongation within 7 days of study day 1 is not permitted unless approved by the sponsor; use of ondansetron is permitted for treatment of nausea and vomiting
* Patients may not be on warfarin, factor Xa inhibitors and direct thrombin inhibitors; Note: low molecular weight heparin and prophylactic low dose warfarin are permitted; APTT/PTT must meet the inclusion criteria; subjects taking low dose warfarin must have their international normalized ratio (INR) followed closely
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible; patients with active infection requiring intravenous (IV) antibiotics within 2 weeks of study day 1 are excluded; patients with myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association [NYHA] class III and higher), unstable angina, or cardiac arrhythmia requiring medication are excluded
* Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis), are ineligible
* Patients with history of bleeding diathesis are ineligible
* Patients with positive hepatitis B surface antigen (HepBsAg), positive hepatitis total core antibody with negative HBsAG, or detectable hepatitis C virus ribonucleic acid (RNA) by a polymerase-chain reaction (PCR) assay are ineligible (screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive)
* Pregnant women are excluded from this study as no studies evaluating the reproductive toxicity of AMG 232 (KRT 232) have been conducted to date; the teratogenic potential of AMG 232 (KRT 232) in laboratory animals, if any, is unknown; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AMG 232 (KRT 232), breastfeeding should be discontinued if the mother is treated with AMG 232 (KRT 232) through 1 week after receiving the last dose of study drug
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AMG 232 (KRT 232); in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients with a planned use of Novo-TTF (Optune) are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameters with target inter-tumor drug concentration at >= 25 nm (Part 1) | Up to 5 years
  Part 2 of the trial will proceed only if at least one of the doses yielded a 50% PK response rate. If both doses reached 50% PK response rate, both doses will be studied in Part 2 of the trial.
Maximum tolerated dose (MTD) of MDM2 inhibitor AMG 232 (KRT-232) when combined with concomitant radiation therapy (Part 2) | Up to 16 weeks
  MTD will be determined according to dose-limiting toxicities graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Beginning April 1, 2018 version 5.0 will be utilized for adverse event reporting). The target dose-limiting toxicity (DLT) rate is 33%. If the MTD is not reached among the pre-specified doses, the dose for the expanded cohort will be the highest dose studied for which the DLT rate is less than 33%.

SECONDARY OUTCOMES:
Incidence of adverse events (Part 1) | Up to 30 days following the last dose of study drug
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Beginning April 1, 2018 version 5.0 will be utilized for adverse event reporting). Will be used for scoring toxicity and adverse events. The severity and frequency of toxicity will be tabulated by the tested dose or doses, or combination regimens using descriptive statistics. The proportion of patients who experienced grade 3 or above toxicities will be estimated along with 95% confidence intervals by each type of toxicity.
Variability of MDM2 inhibitor AMG 232 (KRT-232) concentration in tumor enhancing versus infiltrative tissue (Part 1) | Up to 5 years
  Will be summarized using descriptive statistics.
p21 elevation in tissue (Part 1) | Up to 5 years
  Will be coded as binary outcome either elevated or not elevated compared to a reference value from archived tumor tissues in matched patient population. A proportion of patients with elevated p21 will be estimated using a binomial distribution along with 95% confidence interval.
Incidence of adverse events (Part 2) | Up to 10 weeks
  Assessed by CTCAE version 4.0 (Beginning April 1, 2018 version 5.0 will be utilized for adverse event reporting). Will be used for scoring toxicity and adverse events. The severity and frequency of toxicity will be tabulated by the tested dose or doses, or combination regimens using descriptive statistics. The proportion of patients who experienced grade 3 or above toxicities will be estimated along with 95% confidence intervals by each type of toxicity.
MIC-1 elevation in serum (Part 2) | Up to 5 years
  The PK variables and changes in MIC-1 will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters and MIC-1 changes will be compared across dose level using non-parametric statistical testing techniques.
MDM2 inhibitor AMG 232 (KRT-232) exposure (Part 2) | Up to 5 years
  Assessed by liquid chromatography/tandem mass spectrometry. A full pharmacokinetic profile of AMG 232 (KRT 232) will be proposed in this study to assess exposure-response relationships with various pharmacodynamic (PD) endpoints (i.e., MIC-1 changes, toxicity, and efficacy). Correlation with PD effect on p21 elevation will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Lee, Principal Investigator — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT03107780/ICF_000.pdf